CLINICAL TRIAL: NCT00192985
Title: Does a Nitrofurazone Coated Bladder Catheter Reduce the Number of Urinary Tract Infections in Trauma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: KF 01-160/02 Catheter
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2005-09-19 (Estimated); Status verified 2005-09

CONDITIONS: Trauma; Urinary Tract Infections
MeSH Terms: conditions — Wounds and Injuries; Urinary Tract Infections

INTERVENTIONS:
Device: Nitrofuranzone coated bladder catheter

SUMMARY:
Urinary tract infections occurs in trauma. We investigate whether a nitrofurazone coated can reduce the number of urinary tract infections.

DETAILED DESCRIPTION:
Urinary tract infection occurs in one in five patients as a complication following severe trauma. A new and approved urinary bladder catheter (Releen NF) has been introduced by the Danish company Coloplast A/S. Releen NF is expected to reduce the number of urinary tract infections, but this effect has not been investigated in trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of multiple trauma
* Age >/= 18 years
* Direct referral from scene of accident
* Indication for urinary bladder catherization

Exclusion Criteria:

* Major burn injury
* HIV positiv
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216
Dates: Start 2003-05; Study Completion 2006-09

PRIMARY OUTCOMES:
urinary tract infections

SECONDARY OUTCOMES:
length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Stensballe, MD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Stensballe J, Tvede M, Looms D, Lippert FK, Dahl B, Tonnesen E, Rasmussen LS. Infection risk with nitrofurazone-impregnated urinary catheters in trauma patients: a randomized trial. Ann Intern Med. 2007 Sep 4;147(5):285-93. doi: 10.7326/0003-4819-147-5-200709040-00002. PMID 17785483